CLINICAL TRIAL: NCT02027623
Title: Spinal Control During Functional Activities to Improve Low Back Pain Outcomes
Acronym: LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Linda Van Dillen, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201205051; 2R01HD047709 (NIH)
Record Dates: First submitted 2014-01-02; First posted 2014-01-06 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Mechanical Low Back Pain; Chronic Low Back Pain
Keywords: Mechanical low back pain; Non-specific low back pain; Exercise; Motor skill training
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motor skill training (Experimental): The motor skill training condition involves supervised, massed practice of novel, challenging functional activities that are difficult or painful for the participant to perform due to his low back pain.
  Interventions: Behavioral: Motor skill training
- Strength and flexibility exercise (Active Comparator): The strength and flexibility exercise condition involves performance of 1) strengthening exercises that target all trunk muscles, and 2) flexibility exercises that target all trunk and lower extremity motions.
  Interventions: Behavioral: Strength and flexibility exercise

INTERVENTIONS:
Behavioral: Motor skill training — The participant will assist in selecting both simple and complex functional activities to practice. Difficulty will be graded to match the participant's motor capabilities. Three activities will be practiced per session. Within the practice of activities the training will emphasize 1) contraction of groups of specific trunk muscles, 2) earlier and greater movement of the hip, knee, and/or thoracic spine relative to the lumbar spine, 3) later and less movement of the lumbar spine relative to other regions. Within each activity the conditions of practice will vary based on 1) the participant's ability to perform the activity, and 2) the level of challenge the participant is faced with when performing the activity during his day. Equipment will be provided as needed.
  Arms: Motor skill training
Behavioral: Strength and flexibility exercise — Exercises based on best evidence for effectiveness in people with chronic low back pain will be prescribed. Strengthening exercises will target all trunk muscles. Flexibility exercises will target all trunk and hip motions. All exercises will be performed at the intensity appropriate for the person's musculoskeletal fitness level based on the American College of Sports Medicine guidelines. Difficulty level, frequency, and number of repetitions will be modified based on guidelines described in the literature. Equipment will be provided as needed.
  Arms: Strength and flexibility exercise

SUMMARY:
Exercise is one of the primary interventions used with people with chronic, mechanical low back pain. It is unknown, however, which exercise is best for which person, which exercises a person will adhere to and for how long, and the effect of adhering to a specific type of exercise on how the person functions, particularly in the long run. The purpose of this study is to examine if the short- and long-term effects are different between 1) commonly prescribed strength and flexibility exercises for the trunk and limbs, and 2) individualized practice in daily functional activities that are difficult or painful to perform. Adherence to the different interventions, the relationship between adherence and outcomes,as well as the effect of a booster intervention also will be examined.

DETAILED DESCRIPTION:
For many people, mechanical low back pain (LBP) is a long-term, function-limiting condition rather than a short-term, self-limiting condition. Exercise is one of the primary non-surgical approaches used worldwide for managing LBP. Specifically in people with chronic LBP, exercise has been found to be as efficacious, if not more efficacious than 1) no treatment, 2) usual care, and 3) many other treatments, such as massage or laser therapy. Despite the growing body of evidence for the beneficial effects of exercise, however, there is limited evidence about 1) which exercise is best for which person, 2) how long the effects of different exercises last, 3) which types of exercise people will adhere to, and for how long, and 4) the mechanisms underlying the effects of different types of exercise.

This study aims to address these limitations by directly comparing the effects of 1) exercise to increase strength of the trunk and increase flexibility of the trunk and extremities, and 2) individualized, motor skill training directed at performance of daily functional activities that are painful or limited due to the person's LBP. This study also will examine 1) the effects of a booster phase of intervention, 2) the relationship between adherence to intervention and function, and 3) the relationship between performance of functional activities and function-related outcomes. People with chronic LBP will be randomized to 1) an intervention of strength and flexibility exercise or motor skill training, and 2) a booster or no-booster intervention. Intervention will be provided in 2 phases: 1) initial phase: 6 - 1 hour sessions, once/week for 6 weeks, and 2) booster phase: # of sessions needed to regain independence in home program, beginning 6 months after the initial phase. The investigators will collect 1) measurements of pain, function, disability, and economic outcomes, 2) reports of adherence, and 3) laboratory-based measures of performance of functional activities. People will be followed for 12 months after the initial intervention phase. Three sets of hypotheses are proposed. First, the investigators hypothesize that both interventions will result in improvements in pain, function, disability, and economic outcomes, but that the motor skill training will result in more long lasting improvements than the strength and flexibility exercise. Second, the investigators hypothesize that the effect of a booster phase of intervention will 1) result in longer lasting improvement in function and better adherence than a no-booster intervention, and 2) be greater for motor skill training than for strength and flexibility exercise. Finally, the investigators hypothesize that 1) adherence to motor skill training will be more strongly related to function than will adherence to strength and flexibility exercise, and 2) performance of functional activities by people receiving motor skill training will be more strongly related to function than performance of functional activities by people receiving strength and flexibility exercise.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain for a minimum of 12 months
* currently experiencing low back pain symptoms but not in a recurrence or an acute flare-up
* Modified Oswestry Disability Index score of ≥ 20%
* 3 or more functional activities limited due to low back pain
* able to stand and walk without assistance
* able to understand and sign a consent form

Exclusion Criteria:

* BMI >30
* any structural spinal deformity including scoliosis, kyphosis, or stenosis
* spinal fracture or dislocation
* low back pain due to trauma
* osteoporosis
* ankylosing spondylitis
* rheumatoid arthritis
* fibromyalgia
* symptomatic disc herniation
* spondylolisthesis
* serious spinal complications such as tumor or infection
* previous spinal surgery
* frank neurological loss, i.e., weakness and sensory loss
* pain or paresthesia below the knee
* etiology of low back pain other than the lumbar spine, e.g., hip joint
* history of neurologic disease which required hospitalization
* active treatment for cancer
* history of unresolved cancer
* pregnancy
* worker's compensation, disability, or litigation case
* Graves' disease
* Marfan syndrome
* Unable to classify low back pain based on clinical examination findings

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2014-01-15 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda R Van Dillen, P.T., Ph.D., Principal Investigator — Program in Physical Therapy, Washington University Medical School
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lanier VM, Lohse KR, Hooker QL, Francois SJ, van Dillen LR. Treatment preference changes after exposure to treatment in adults with chronic low back pain. PM R. 2023 Jul;15(7):817-827. doi: 10.1002/pmrj.12897. Epub 2022 Oct 24. PMID 36106673
- [Derived] van Dillen LR, Lanier VM, Steger-May K, Wallendorf M, Norton BJ, Civello JM, Czuppon SL, Francois SJ, Roles K, Lang CE. Effect of Motor Skill Training in Functional Activities vs Strength and Flexibility Exercise on Function in People With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Neurol. 2021 Apr 1;78(4):385-395. doi: 10.1001/jamaneurol.2020.4821. PMID 33369625
- [Derived] Francois SJ, Lanier VM, Marich AV, Wallendorf M, Van Dillen LR. A Cross-Sectional Study Assessing Treatment Preference of People With Chronic Low Back Pain. Arch Phys Med Rehabil. 2018 Dec;99(12):2496-2503. doi: 10.1016/j.apmr.2018.04.027. Epub 2018 May 28. PMID 29852151

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was by way of flyers placed in the community and physician offices, ads and interviews through local media and clinics in the region. Recruitment spanned December 2013 to August 2016.
Groups:
- Motor Skill Training: The motor skill training condition involves supervised, massed practice of novel, challenging functional activities that are difficult or painful for the participant to perform due to his low back pain.
  Motor skill training: The participant will assist in selecting both simple and complex functional activities to practice. Difficulty will be graded to match the participant's motor capabilities. Three activities will be practiced per session. Within the practice of activities the training will emphasize 1) contraction of groups of specific trunk muscles, 2) earlier and greater movement of the hip, knee, and/or thoracic spine relative to the lumbar spine, 3) later and less movement of the lumbar spine relative to other regions. Within each activity the conditions of practice will vary based on 1) the participant's ability to perform the activity, and 2) the level of challenge the participant is faced with when performing the activity during his day. Equipment provided as needed.
Period: Overall Study
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Started | 77 | 77
Completed | 68 | 65
Not Completed | 9 | 12
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 6 | 9

BASELINE CHARACTERISTICS:
Population: N=149; five participants (3=MST, 2=SF) excluded from analysis due to only have a baseline time point.
Groups:
- Total: Total of all reporting groups
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise | Total
Number analyzed (Participants) | 74 | 75 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (11.8) | 42.6 (11.7) | 42.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 41 | 91
  Male | 24 | 34 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 12 | 11 | 23
  White | 54 | 56 | 110
  More than one race | 5 | 1 | 6
  Unknown or Not Reported | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.3 (3.2) | 26.1 (3.1) | 25.7 (3.2)
Married or living with significant other [Count of Participants; unit: Participants] | 45 | 55 | 100
Completed at least some college [Count of Participants; unit: Participants] | 67 | 72 | 139
Employment situation [Count of Participants; unit: Participants]
  Working full-time | 50 | 51 | 101
  Working part-time | 15 | 13 | 28
  Student (not working) | 4 | 1 | 5
  Other employment status | 5 | 10 | 15
Low Back Pain Classification [Count of Participants; unit: Participants]
  Rotation | 42 | 40 | 82
  Rotation with flexion | 1 | 3 | 4
  Rotation with extension | 31 | 32 | 63
Duration of Low Back Pain [Median (Inter-Quartile Range); unit: years] | 7.0 [3 to 20] | 7.0 [4 to 15] | 7.0 [3 to 15]
Symptoms only in the back [Count of Participants; unit: Participants] | 58 | 54 | 112
Fear-Avoidance Beliefs Questionnaire - Physical Activity Subscale Score [Mean (Standard Deviation); unit: units on a scale] — Assess a participant's fear of pain and beliefs about how physical activity affects his low back pain. The physical activity subscale score ranges from 0-24 with higher scores indicating higher fear-avoidance beliefs about physical activity.
  units on a scale | 14.7 (6.1) | 14.1 (5.1) | 14.4 (5.6)
Fear-Avoidance Beliefs Questionnaire - Work Subscale Score [Mean (Standard Deviation); unit: units on a scale] — Assess a participant's fear of pain and beliefs about how work affects his low back pain. The work subscale score ranges from 0-42 with higher scores indicating higher fear-avoidance beliefs about work.
  units on a scale | 10.9 (8.4) | 11.8 (9.0) | 11.4 (8.7)
Modified Oswestry Disability Questionnaire [Mean (Standard Deviation); unit: units on a scale] — A disease-specific measure that provides an index of a participant's perceived low back pain-related functional limitation. The scale for the Modified Oswestry Disability Questionnaire ranges from 0-100; 100 represents the highest level of limitation.
  units on a scale | 32.3 (10.2) | 32.6 (9.4) | 32.4 (9.8)
NRS average pain prior 7 days [Mean (Standard Deviation); unit: units on a scale] — Numeric Pain Rating Scale of average pain in the prior 7 days: An 11-point scale (0-10) where participants rate their average low back pain symptoms in the prior 7 days on a numeric scale of 0-10 where 0 represents no symptoms and 10 represents symptoms as bad as can be.
  units on a scale | 4.7 (1.9) | 4.7 (1.5) | 4.7 (1.7)
NRS worst pain, prior 7 days [Mean (Standard Deviation); unit: units on a scale] — Numeric Pain Rating Scale of worst pain in the prior 7 days: An 11-point scale (0-10) where participants rate their worst low back pain symptoms in the prior 7 days on a numeric scale of 0-10 where 0 represents no symptoms and 10 represents symptoms as bad as can be.
  units on a scale | 6.3 (2) | 6.9 (1.6) | 6.6 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Modified Oswestry Disability Questionnaire (0-100%) From Baseline to Completion of Initial 6 Week Intervention Phase
Description: Background/Purpose: The 10-item Modified Oswestry Disability Questionnaire is a disease-specific measure that provides an index of a participant's perceived low back pain-related functional limitation.
  Procedure: Participants will answer each of the 10 questions by placing a mark in the one box that best describes his current condition. Since a participant may feel that 2 of the statements describe his condition, he is instructed to mark only the box that most closely describes his current condition.
  Scoring: Each item is given a value from 0-5. The total score is the sum of all questions divided by 50, multiplied by 100 to get a percent. 100 represents the highest level of limitation.
Time Frame: Baseline, completion of initial 6 week intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 74 | 75
score on a scale
  Baseline | 32.3 (10.2) | 32.6 (9.4)
  Post-Treatment: number analyzed (Participants) | 68 | 67
  Post-Treatment | 12.8 (10.7) | 21.2 (10.7)

2. Primary Outcome: Change in Modified Oswestry Disability Questionnaire (0-100%) From Completion of Initial 6 Week Intervention Phase to 6 Months After Initial Intervention Phase
Description: as for outcome 1
Time Frame: Completion of initial 6 week intervention phase, 6 months after initial intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 68 | 67
score on a scale
  Post-Treatment | 12.8 (10.7) | 21.2 (10.7)
  Follow-Up Month 6 | 12.0 (12.6) | 18.2 (10.5)

3. Primary Outcome: Change in Modified Oswestry Disability Questionnaire (0-100%) From 6 Months After Initial Intervention Phase to 12 Months After Initial Intervention Phase
Description: as for outcome 1
Time Frame: 6 months after initial intervention phase, 12 months after initial intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 68 | 67
score on a scale
  Follow-Up Month 6 | 12.0 (12.6) | 18.2 (10.5)
  Follow-Up Month 12: number analyzed (Participants) | 68 | 65
  Follow-Up Month 12 | 10.8 (11.3) | 16.7 (11.3)

4. Secondary Outcome: Change in Numeric Pain Rating Scale (0-10) From Baseline to Completion of Initial 6 Week Intervention Phase
Description: Background/Purpose: This questionnaire is designed to give the therapist information on the intensity of a participant's LBP symptoms.
  Procedure: Participants will rate their LBP symptoms on a numeric scale of 0-10 where 0 represents no symptoms and 10 represents symptoms as bad as can be. They will rate their average symptoms over the prior 7 days, and worst symptoms over the prior 7 days.
  Scoring: The score for each item is the rating the participant provides for each symptom category (average and worst).
Time Frame: Baseline, completion of initial 6 week intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 74 | 75
units on a scale
  Baseline (Average) | 4.7 (1.9) | 4.7 (1.5)
  Post-Treatment (Average): number analyzed (Participants) | 68 | 67
  Post-Treatment (Average) | 1.4 (1.1) | 2.1 (1.2)
  Baseline (Worst) | 6.3 (2.0) | 6.9 (1.6)
  Post-Treatment (Worst): number analyzed (Participants) | 68 | 67
  Post-Treatment (Worst) | 2.7 (1.7) | 4.0 (1.9)

5. Secondary Outcome: Change in Numeric Pain Rating Scale (0-10) From Completion of Initial 6 Week Intervention Phase to 6 Months After Initial Intervention Phase
Description: as for outcome 4
Time Frame: Completion of initial 6 week intervention phase, 6 months after initial intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 68 | 67
units on a scale
  Post-Treatment (Average) | 1.4 (1.1) | 2.1 (1.2)
  Follow-Up Month 6 (Average) | 2.0 (1.8) | 2.6 (1.8)
  Post-Treatment (Worst) | 2.7 (1.7) | 4.0 (1.9)
  Follow-Up Month 6 (Worst) | 2.9 (2.2) | 3.8 (2.2)

6. Secondary Outcome: Change in Numeric Pain Rating Scale (0-10) From 6 Months After Initial Intervention Phase to 12 Months After Initial Intervention Phase
Description: as for outcome 4
Time Frame: 6 months after initial intervention phase, 12 months after initial intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 68 | 67
units on a scale
  Follow-Up Month 6 (Average) | 2.0 (1.8) | 2.6 (1.8)
  Follow-Up Month 12 (Average): number analyzed (Participants) | 68 | 65
  Follow-Up Month 12 (Average) | 1.8 (1.9) | 2.6 (2.0)
  Follow-Up Month 6 (Worst) | 2.9 (2.2) | 3.8 (2.2)
  Follow-Up Month 12 (Worst): number analyzed (Participants) | 68 | 65
  Follow-Up Month 12 (Worst) | 2.8 (2.3) | 3.9 (2.5)

7. Secondary Outcome: Change in Number of Acute Flare-ups of Low Back Pain (#) in Past 6 Months, From Baseline to 6 Months After Initial Intervention Phase
Description: Background/Purpose: This questionnaire is designed to give the therapist information about the history of a participant's LBP flare-ups in the past 6 months.
  Definition: A flare-up is an increase in symptoms of at least 2 points on the NRS above a person's typical low back pain and lasts for at least 2 consecutive days Procedure: Participants will fill in information on how many acute flare-ups they have had over the past 6 months.
  Scoring: The score will be the number the participant provides for the number of acute flare-ups over the last 6 months.
Time Frame: Baseline, 6 months after initial intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: acute flare-ups
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 74 | 75
acute flare-ups
  Baseline | 7.1 (7.6) | 9.8 (11.9)
  Follow-Up Month 6: number analyzed (Participants) | 65 | 60
  Follow-Up Month 6 | 2.0 (3.3) | 4.2 (8.2)

8. Secondary Outcome: Change in Number of Acute Flare-ups of Low Back Pain (#) in Past 6 Months, From 6 Months After the Initial Intervention Phase to 12 Months After Initial Intervention Phase
Description: as for outcome 7
Time Frame: 6 months after initial intervention phase, 12 months after initial intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: acute flare-ups
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 67 | 64
acute flare-ups
  Follow-Up Month 6: number analyzed (Participants) | 65 | 60
  Follow-Up Month 6 | 2.0 (3.3) | 4.2 (8.2)
  Follow-Up Month 12 | 1.3 (1.8) | 2.0 (2.8)

9. Secondary Outcome: Change in Current Medication Use for Low Back Pain (Number of Participants Currently Using Medication) From Baseline to Completion of Initial 6 Week Intervention Phase
Description: Background/Purpose: This questionnaire is designed to provide general information on the use of medication for a participant's LBP.
  Procedure: Participants will answer each question by marking if they are taking non-prescription medication and prescription medication for their LBP. Reported as number of participants currently using medication for LBP.
Time Frame: Baseline, completion of initial 6 week intervention phase
Population: Data available at the time points
Measure: Count of Participants; unit: Participants
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 74 | 75
Participants
  Baseline | 50 | 47
  Post-Treatment: number analyzed (Participants) | 70 | 67
  Post-Treatment | 21 | 31

10. Secondary Outcome: Change in Current Medication Use for Low Back Pain (Number of Participants Currently Using Medication) From Completion of Initial 6 Week Intervention Phase to 6 Months After Initial Intervention Phase
Description: as for outcome 9
Time Frame: Completion of initial 6 week intervention phase, 6 months after initial intervention phase
Population: Data available at the time points
Measure: Count of Participants; unit: Participants
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 70 | 67
Participants
  Post-Treatment | 21 | 31
  Follow-Up Month 6: number analyzed (Participants) | 68 | 62
  Follow-Up Month 6 | 27 | 29

11. Secondary Outcome: Change in Current Medication Use for Low Back Pain (Number of Participants Currently Using Medication) From 6 Months After Completion of Initial Intervention Phase to 12 Months After Completion of Initial Intervention Phase
Description: as for outcome 9
Time Frame: 6 months after initial intervention phase, 12 months after initial intervention phase
Population: Data available at the time points
Measure: Count of Participants; unit: Participants
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 68 | 66
Participants
  Follow-Up Month 6: number analyzed (Participants) | 68 | 62
  Follow-Up Month 6 | 27 | 29
  Follow-Up Month 12 | 23 | 25

12. Secondary Outcome: Change in Absenteeism From Usual Activities Due to Low Back Pain (Number of Participants Who Report Absenteeism) From Baseline to Completion of Initial 6 Week Intervention Phase
Description: Background/Purpose: This questionnaire is designed to assess the number of days a participant has been kept from his usual activities (work, school or housework) because of LBP.
  Procedure: Participants will answer each question by marking the answer as indicated.
  Scoring: Reported as the number of participants who reported absenteeism from usual activities over the past 4 weeks.
Time Frame: Baseline, completion of initial 6 week intervention phase
Population: Data available at the time points
Measure: Count of Participants; unit: Participants
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 74 | 75
Participants
  Baseline | 42 | 47
  Post-Treatment: number analyzed (Participants) | 68 | 67
  Post-Treatment | 11 | 29

13. Secondary Outcome: Change in Absenteeism From Usual Activities Due to Low Back Pain (Number of Participants Who Report Absenteeism) From Completion of Initial 6 Week Intervention Phase to 6 Months After Initial Intervention Phase
Description: as for outcome 12
Time Frame: Completion of initial 6 week intervention phase, 6 months after initial intervention phase
Population: Data available at the time points
Measure: Count of Participants; unit: Participants
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 68 | 67
Participants
  Post-Treatment | 11 | 29
  Follow-Up Month 6 | 9 | 11

14. Secondary Outcome: Change in Absenteeism From Usual Activities Due to Low Back Pain (Number of Participants Who Report Absenteeism) From 6 Months After Initial Intervention Phase to 12 Months After Initial Intervention Phase
Description: as for outcome 12
Time Frame: 6 months after initial intervention phase, 12 months after initial intervention phase
Population: Data available at the time points
Measure: Count of Participants; unit: Participants
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 68 | 67
Participants
  Follow-Up Month 6 | 9 | 11
  Follow-Up Month 12: number analyzed (Participants) | 68 | 65
  Follow-Up Month 12 | 11 | 12

15. Secondary Outcome: Change in Stanford Presenteeism Scale (Work Impairment Score: 10-50) From Baseline to Completion of Initial 6 Week Intervention Phase
Description: Background/Purpose: This questionnaire is designed to assess how a participant's LBP affected his participation in usual activities and the impact of LBP on his ability to do his job over the past 4 weeks.
  Scoring: A Work Impairment Score (WIS) is calculated as the sum of answers on the questions regarding how LBP has affected job ability over the past 4 weeks. Each of the WIS questions is ranked on a 5-point Likert scale. All scores are 1-5, with questions 2, 5, 6, 8, and 10 reverse scored (5-1). The score ranges from 10-50 with 50 indicating the highest degree of impairment.
Time Frame: Baseline, completion of initial 6 week intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline | 20.3 (5.3) | 19.9 (6.2)
  Post-Treatment: number analyzed (Participants) | 57 | 55
  Post-Treatment | 17.4 (4.6) | 18.3 (5.2)

16. Secondary Outcome: Change in Stanford Presenteeism Scale (Work Impairment Score: 10-50) From Completion of Initial 6 Week Intervention Phase to 6 Months After Initial Intervention Phase
Description: as for outcome 15
Time Frame: Completion of initial 6 week intervention phase, 6 months after initial intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 59 | 59
score on a scale
  Post-Treatment: number analyzed (Participants) | 57 | 55
  Post-Treatment | 17.4 (4.6) | 18.3 (5.2)
  Follow-Up Month 6 | 15.9 (5.6) | 16.5 (5.3)

17. Secondary Outcome: Change in Stanford Presenteeism Scale (Work Impairment Score: 10-50) From 6 Months After Initial Intervention Phase to 12 Months After Initial Intervention Phase
Description: as for outcome 15
Time Frame: 6 months after initial intervention phase, 12 months after initial intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 59 | 59
score on a scale
  Follow-Up Month 6 | 15.9 (5.6) | 16.5 (5.3)
  Follow-Up Month 12: number analyzed (Participants) | 58 | 56
  Follow-Up Month 12 | 15.4 (5.1) | 16.7 (6.0)

18. Secondary Outcome: Change in 36-Item Short Form Health Survey (SF-36) Physical Component Summary Score From Baseline to Completion of Initial 6 Week Intervention Phase
Description: Background/Purpose: This questionnaire is designed to assess information about a participant's mental and physical health, and how well he is able to do his usual activities.
  Procedure: Participants will answer each question by marking the answer as indicated. If participants are unsure how to answer a question, they are instructed to choose the best answer they can.
  Scoring: Using a scoring application, the SF-36 provides 8 scales: a Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and a Mental Health score. The scores are combined to provide a Physical Component (PCS) and Mental Component (MCS) Summary score. For the PCS and the MCS, norm-based scores are scaled and normalized to have a mean of 50 and a standard deviation of 10 based on the 1998 population norms. Higher scores indicate better health.
Time Frame: Baseline, completion of initial 6 week intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 74 | 75
T-scores
  Baseline | 43.2 (6.6) | 40.8 (6.9)
  Post-Treatment: number analyzed (Participants) | 68 | 67
  Post-Treatment | 50.8 (6.5) | 46.3 (7.0)

19. Secondary Outcome: Change in 36-Item Short Form Health Survey (SF-36) Physical Component Summary Score From Completion of Initial 6 Week Intervention Phase to 6 Months After Initial Intervention Phase
Description: as for outcome 18
Time Frame: Completion of initial 6 week intervention phase, 6 months after initial intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 68 | 67
T-scores
  Post-Treatment | 50.8 (6.5) | 46.3 (7.0)
  Follow-Up Month 6: number analyzed (Participants) | 65 | 60
  Follow-Up Month 6 | 50.9 (6.6) | 47.8 (7.4)

20. Secondary Outcome: Change in 36-Item Short Form Health Survey (SF-36) Physical Component Summary Score From 6 Months After Initial Intervention Phase to 12 Months After Initial Intervention Phase
Description: as for outcome 18
Time Frame: 6 months after initial intervention phase, 12 months after initial intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 66 | 64
T-scores
  Follow-Up Month 6: number analyzed (Participants) | 65 | 60
  Follow-Up Month 6 | 50.9 (6.6) | 47.8 (7.4)
  Follow-Up Month 12 | 51.2 (8.0) | 48.3 (7.4)

21. Secondary Outcome: Change in 36-Item Short Form Health Survey (SF-36) Mental Component Summary Score From Baseline to Completion of Initial 6 Week Intervention Phase
Description: as for outcome 18
Time Frame: Baseline, completion of initial 6 week intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 74 | 75
T-scores
  Baseline | 49.2 (11.6) | 52.1 (9.3)
  Post-Treatment: number analyzed (Participants) | 68 | 67
  Post-Treatment | 50.7 (8.6) | 51.0 (11.6)

22. Secondary Outcome: Change in 36-Item Short Form Health Survey (SF-36) Mental Component Summary Score From Completion of Initial 6 Week Intervention Phase to 6 Months After Initial Intervention Phase
Description: as for outcome 18
Time Frame: Completion of initial 6 week intervention phase, 6 months after initial intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 68 | 67
T-scores
  Post-Treatment | 50.7 (8.6) | 51.0 (11.6)
  Follow-Up Month 6: number analyzed (Participants) | 65 | 60
  Follow-Up Month 6 | 49.6 (10.5) | 50.8 (10.4)

23. Secondary Outcome: Change in 36-Item Short Form Health Survey (SF-36) Mental Component Summary Score From 6 Months After Initial Intervention Phase to 12 Months After Initial Intervention Phase
Description: as for outcome 18
Time Frame: 6 months after initial intervention phase, 12 months after initial intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 66 | 64
T-scores
  Follow-Up Month 6: number analyzed (Participants) | 65 | 60
  Follow-Up Month 6 | 49.6 (10.5) | 50.8 (10.4)
  Follow-Up Month 12 | 50.4 (10.3) | 50.3 (11.5)

24. Secondary Outcome: Change in Use of Other Low Back Pain-related Treatments (Health Professional Care Seeking or Equipment Use (# of Participants)) From Baseline to Completion of Initial 6 Week Intervention Phase
Description: Background/Purpose: This questionnaire is designed to provide general information on the use of additional treatments for a participant's LBP.
  Health Professional Care Seeking Procedure: Participants will answer each question by marking yes or no for a list of other healthcare professionals they are seeing for treatment of their LBP.
  Equipment Use Procedure: Participants will answer each question by marking yes or no for a list of equipment they are using to treat their LBP.
  Scoring: Reported as the number of participants seeking care from health professionals for LBP or using equipment for LBP.
Time Frame: Baseline, completion of initial 6 week intervention phase
Population: Data available at the time points
Measure: Count of Participants; unit: Participants
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 74 | 75
Participants
  Baseline (Care Seeking) | 35 | 29
  Post-Treatment (Care Seeking): number analyzed (Participants) | 68 | 67
  Post-Treatment (Care Seeking) | 7 | 6
  Baseline (Equipment Use) | 66 | 65
  Post-Treatment (Equipment Use): number analyzed (Participants) | 68 | 67
  Post-Treatment (Equipment Use) | 62 | 48

25. Secondary Outcome: Change in Use of Other Low Back Pain-related Treatments (Health Professional Care Seeking or Equipment Use (# of Participants)) From Completion of Initial 6 Week Intervention Phase to 6 Months After Initial Intervention Phase
Description: as for outcome 24
Time Frame: Completion of initial 6 week intervention phase, 6 months after initial intervention phase
Population: Data available at the time points
Measure: Count of Participants; unit: Participants
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 68 | 67
Participants
  Post-Treatment (Care Seeking) | 7 | 6
  Follow-Up Month 6 (Care Seeking) | 13 | 13
  Post-Treatment (Equipment Use) | 62 | 48
  Follow-Up Month 6 (Equipment Use) | 33 | 29

26. Secondary Outcome: Change in Use of Other Low Back Pain-related Treatments (Health Professional Care Seeking or Equipment Use (# of Participants)) From 6 Months After Initial Intervention Phase to 12 Months After Initial Intervention Phase
Description: as for outcome 24
Time Frame: 6 months after initial intervention phase, 12 months after initial intervention phase
Population: Data available at the time points
Measure: Count of Participants; unit: Participants
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 68 | 67
Participants
  Follow-Up Month 6 (care seeking) | 13 | 13
  Follow-Up Month 12 (care seeking): number analyzed (Participants) | 68 | 65
  Follow-Up Month 12 (care seeking) | 8 | 11
  Follow-Up Month 6 (equipment use) | 33 | 29
  Follow-Up Month 12 (equipment use): number analyzed (Participants) | 68 | 65
  Follow-Up Month 12 (equipment use) | 28 | 30

27. Secondary Outcome: Satisfaction With Care (15-75 Points)
Description: Background/Purpose: This questionnaire assesses information about how satisfied a participant feels with the physical therapist and treatment he was provided.
  Procedure: Participants will answer each question by marking the answer as indicated. They may only check off one answer per item.
  Scoring: Each question is ranked on a 5-point Likert scale. All scores are 1-5, with questions 1, 3, 4, 8, 9, 10 and 13 reverse scored (5-1). The total score is the sum of all of the answers (15-75) with higher scores indicating more satisfaction with care.
Time Frame: Completion of initial 6 week intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 68 | 67
score on a scale | 68.8 (0.9) | 61.4 (0.9)

28. Secondary Outcome: Change in Kinematics During Functional Activities (Degrees) From Baseline to Completion of Initial 6 Week Intervention Phase
Description: Background/Purpose: These are laboratory measures of (1) movement of the lumbar region, hips and knees or (2) static alignment of the lumbar region during functional activities. Procedures: Angular data is quantified based on data from retro-reflective markers that are tracked with a 3-dimensional video system while the person performs an activity. Coordinate data from the video system is processed to provide quantification of movement or alignment. The variables of interest are (1) angular excursion in the first 50% of the descent phase for each region or joint during picking up an object and (2) lumbar curvature angle for preferred sitting. For movement, smaller numbers from baseline to post-treatment represent decreased movement of a region or joint. For alignment, larger negative numbers from baseline to post-treatment represent a more extended lumbar region alignment. Measures are obtained at baseline and immediately after a 6-week intervention phase.
Time Frame: Baseline, completion of initial 6 week intervention phase
Population: Data available at the time points
Measure: Mean (95% Confidence Interval); unit: Angle in degrees
Groups:
- Motor Skill Training: The motor skill training condition involves supervised, massed practice of novel, challenging functional activities that are difficult or painful for the participant to perform due to his low back pain.
  Motor skill training: The participant will assist in selecting both simple and complex functional activities to practice. Difficulty will be graded to match the participant's capabilities. Three activities will be practiced per session. Within the practice of activities the training will emphasize 1) contraction of groups of specific trunk muscles, 2) earlier and greater movement of the hip, knee, and/or thoracic spine relative to the lumbar spine, 3) later and less movement of the lumbar spine relative to other regions. The conditions of practice will vary based on 1) ability to perform the activity, and 2)level of challenge the participant is faced with performing the activity during his day. Equipment will be provided as needed.
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 76 | 77
Angle in degrees
  Baseline: Lumbar region excursion | 11.32 [10.36 to 12.29] | 11.23 [10.28 to 12.17]
  Post-intervention: Lumbar region: number analyzed (Participants) | 68 | 67
  Post-intervention: Lumbar region | 9.17 [8.33 to 10.00] | 11.05 [9.94 to 12.16]
  Baseline: Hip joint excursion | 21.17 [19.18 to 23.16] | 20.84 [18.78 to 22.90]
  Post-intervention: Hip joint excursion: number analyzed (Participants) | 68 | 67
  Post-intervention: Hip joint excursion | 31.98 [29.84 to 34.13] | 20.36 [18.46 to 22.25]
  Baseline: Knee joint excursion | 11.08 [8.04 to 14.11] | 8.86 [5.81 to 11.90]
  Post-intervention: Knee joint excursion: number analyzed (Participants) | 68 | 67
  Post-intervention: Knee joint excursion | 30.10 [26.96 to 33.25] | 9.69 [6.15 to 13.24]
  Baseline: Lumbar region curvature | -5.91 [-7.91 to -3.88] | -3.18 [-5.09 to -1.27]
  Post-intervention: Lumbar region curvature: number analyzed (Participants) | 67 | 67
  Post-intervention: Lumbar region curvature | -7.51 [-9.70 to -5.33] | -6.45 [-8.52 to -4.38]

29. Secondary Outcome: Change in Kinematics During Functional Activities (Degrees) From Completion of Initial 6 Week Intervention Phase to 6 Months After Intervention Phase
Description: Background/Purpose: These are laboratory measures of (1) movement of the lumbar region, hips and knees or (2) static alignment of the lumbar region during functional activities. Procedures: Angular data is quantified based on data from retro-reflective markers that are tracked with a 3-dimensional video system while the person performs an activity. Coordinate data from the video system is processed to provide quantification of movement or alignment. The variables of interest are (1) angular excursion in the first 50% of the descent phase for each region or joint during picking up an object and (2) lumbar curvature angle for preferred sitting. For movement, smaller numbers from baseline to post-treatment represent decreased movement of a region or joint. For alignment, larger negative numbers from baseline to post-treatment represent a more extended lumbar region alignment. Measures are obtained after a 6 week intervention phase and 6 months after intervention.
Time Frame: Completion of initial 6 week intervention phase, 6 months after initial intervention phase
Population: Data available at the time points
Measure: Mean (95% Confidence Interval); unit: Angle in degrees
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 68 | 67
Angle in degrees
  Post-intervention: Lumbar excursion | 9.17 [8.33 to 10.00] | 11.05 [9.94 to 12.16]
  6 months post-intervention: Lumbar excursion: number analyzed (Participants) | 65 | 60
  6 months post-intervention: Lumbar excursion | 8.63 [7.71 to 9.55] | 10.84 [9.73 to 11.96]
  Post-intervention: Hip joint excursion | 31.98 [29.84 to 34.13] | 20.36 [18.46 to 22.25]
  6 months post-intervention: Hip joint excursion: number analyzed (Participants) | 65 | 60
  6 months post-intervention: Hip joint excursion | 30.03 [27.70 to 32.35] | 20.08 [18.39 to 21.78]
  Post-intervention: Knee joint excursion | 30.10 [26.96 to 33.25] | 9.69 [6.15 to 13.20]
  6 months post intervention: Knee joint excursion: number analyzed (Participants) | 65 | 60
  6 months post intervention: Knee joint excursion | 26.90 [23.83 to 29.97] | 9.81 [6.43 to 13.20]
  Post-intervention: Lumbar curvature: number analyzed (Participants) | 67 | 67
  Post-intervention: Lumbar curvature | -7.51 [-9.70 to -5.33] | -6.45 [-8.52 to -4.38]
  6 months post-intervention: Lumbar curvature: number analyzed (Participants) | 65 | 60
  6 months post-intervention: Lumbar curvature | -5.43 [-7.63 to -3.24] | -5.89 [-7.79 to -3.99]

30. Other Pre Specified Outcome: Adherence to Home Program (0-100%) at Completion of Initial 6 Week Intervention Phase
Description: Background/Purpose: This questionnaire is designed to provide information about how often a participant performs his treatment as it was prescribed.
  Procedure: Participants will use a VAS to indicate for each day the percentage of the treatment they were able to perform as prescribed. At each clinic visit the therapist will ask the participant to provide an estimate of the average percentage of the treatment he was able to perform as prescribed in the interval of time between 2 clinic visits.
  Scoring: Average adherence is calculated by averaging the participants' daily adherence. Scores range from 0-100%. Higher values indicate higher adherence to treatment.
Time Frame: completion of initial 6 week intervention phase
Population: Data available at this time point
Measure: Mean (Standard Deviation); unit: percentage of adherence to home program
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 71 | 72
percentage of adherence to home program | 83 (14) | 90 (15)

31. Other Pre Specified Outcome: Adherence to Home Program (0-100%) at 6 Months After Completion of Initial Intervention Phase
Description: Background/Purpose: This questionnaire is designed to provide information about how often a participant performs his treatment as it was prescribed.
  Procedure: Participants will use a VAS to indicate an average percent adherence to performance of the treatment as prescribed over the past month.
  Scoring: Value (percentage of treatment performed) provided by the participant on each monthly survey. Scores range from 0-100%. Higher values indicate higher adherence to treatment.
Time Frame: 6 months after initial intervention phase
Population: Data available at this time point
Measure: Mean (Standard Deviation); unit: percentage of adherence to home program
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 68 | 67
percentage of adherence to home program | 70 (21) | 42 (31)

32. Other Pre Specified Outcome: Adherence to Home Program (0-100%) at 12 Months After Initial Intervention Phase
Description: as for outcome 31
Time Frame: 12 months after initial intervention phase
Population: Data available at this time point
Measure: Mean (Standard Deviation); unit: percentage of adherence to home program
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 68 | 65
percentage of adherence to home program | 66 (21) | 52 (35)

33. Other Pre Specified Outcome: Change in Fear-Avoidance Beliefs Questionnaire Work Subscale Score (0-42 Points) From Baseline to Completion of Initial 6 Week Intervention Phase
Description: Background/Purpose: This questionnaire is designed to assess a participant's fear of pain and beliefs about how work and physical activity affect his LBP.
  Procedure: Participants will answer each question by marking the answer as indicated.
  Scoring: Each question is ranked on a 7-point Likert scale (0-6). Higher scores indicate higher fear-avoidance. Two subscale scores are calculated. The physical activity subscale score (FABQ-PA) is the sum of questions 2, 3, 4, and 5 and ranges from 0-24. The work subscale score (FABQ-W) is the sum of items 6, 7, 9, 10, 11, 12, and 15 and ranges from 0-42.
Time Frame: Baseline, completion of initial 6 week intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 74 | 75
score on a scale
  Baseline | 10.9 (8.4) | 11.8 (9.0)
  Post-Treatment: number analyzed (Participants) | 68 | 67
  Post-Treatment | 7.7 (7.1) | 10.9 (9.5)

34. Other Pre Specified Outcome: Change in Fear-Avoidance Beliefs Questionnaire Work Subscale Score (0-42 Points) From Completion of Initial 6 Week Intervention Phase to 6 Months After Initial Intervention Phase
Description: as for outcome 33
Time Frame: Completion of initial 6 week intervention phase, 6 months after initial intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 68 | 67
score on a scale
  Post-Treatment | 7.7 (7.1) | 10.9 (9.5)
  Follow-Up Month 6: number analyzed (Participants) | 65 | 60
  Follow-Up Month 6 | 7.2 (8.2) | 9.0 (8.7)

35. Other Pre Specified Outcome: Change in Fear-Avoidance Beliefs Questionnaire Work Subscale Score (0-42 Points) From 6 Months After Initial Intervention Phase to 12 Months After Initial Intervention Phase
Description: as for outcome 33
Time Frame: 6 months after initial intervention phase, 12 months after initial intervention phase
Population: Data for 12 months after the initial intervention phase were not collected. The decision not to collect 12 month data was made prior to finalization of the protocol and participant enrollment.
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 0 | 0

36. Other Pre Specified Outcome: Change in Fear-Avoidance Beliefs Questionnaire Physical Activity Subscale Score (0-24 Points) From Baseline to Completion of Initial 6 Week Intervention Phase
Description: as for outcome 33
Time Frame: Baseline, completion of initial 6 week intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 74 | 75
score on a scale
  Baseline | 14.7 (6.1) | 14.1 (5.1)
  Follow-Up Month 6: number analyzed (Participants) | 68 | 67
  Follow-Up Month 6 | 11.4 (5.9) | 11.6 (5.3)

37. Other Pre Specified Outcome: Change in Fear-Avoidance Beliefs Questionnaire Physical Activity Subscale Score (0-24 Points) From Completion of Initial 6 Week Intervention Phase to 6 Months After Initial Intervention Phase
Description: as for outcome 33
Time Frame: Completion of initial 6 week intervention phase, 6 months after initial intervention phase
Population: Data available at the time points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 68 | 67
score on a scale
  Post-Treatment | 11.4 (5.9) | 11.6 (5.3)
  Follow-Up Month 6: number analyzed (Participants) | 65 | 60
  Follow-Up Month 6 | 11.0 (5.8) | 11.4 (5.5)

38. Other Pre Specified Outcome: Change in Fear-Avoidance Beliefs Questionnaire Physical Activity Subscale Score (0-24 Points) From 6 Months After Initial Intervention Phase to 12 Months After Initial Intervention Phase
Description: as for outcome 33
Time Frame: 6 months after initial intervention phase, 12 months after initial intervention phase
Population: as for outcome 35
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 0 | 0

39. Other Pre Specified Outcome: Treatment Preference Assessment Measure, Effectiveness Subscale (0-4 Points)
Description: Background/Purpose: This questionnaire is designed to provide information about a participant's treatment preferences and the participant's perceptions of four attributes of each treatment: effectiveness, acceptability, suitability/appropriateness, and convenience. The questionnaire is modified from a preference questionnaire designed by Sidani et al to reflect the treatments provided in the trial.
  Procedure: The two treatment descriptions will be given in a random order to each participant.
  Scoring: The four treatment attributes (effectiveness, acceptability, suitability/appropriateness, and convenience) will be rated on a 5-point Likert scale (0-4). The anchors are not at all (rating=0) and very much (rating=4).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 74 | 75
units on a scale
  Effectiveness of Motor Skill Training | 2.28 (1.14) | 2.36 (1.00)
  Effectiveness of Strength and Flexibility Exercise | 3.19 (0.81) | 2.92 (0.82)

40. Other Pre Specified Outcome: Treatment Preference Assessment Measure, Acceptability Subscale (0-4 Points)
Description: as for outcome 39
Time Frame: Baseline
Population: Data available at this time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 74 | 75
units on a scale
  Acceptability of Motor Skill Training: number analyzed (Participants) | 74 | 74
  Acceptability of Motor Skill Training | 2.66 (1.09) | 2.72 (0.97)
  Acceptability of Strength and Flexibility Exercise | 3.37 (0.69) | 3.21 (0.70)

41. Other Pre Specified Outcome: Treatment Preference Assessment Measure, Suitability/Appropriateness Subscale (0-4 Points)
Description: as for outcome 39
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 74 | 75
units on a scale
  Suitability of Motor Skill Training | 2.43 (1.14) | 2.48 (1.20)
  Suitability of Strength and Flexibility Exercise | 3.31 (0.74) | 3.15 (0.80)

42. Other Pre Specified Outcome: Treatment Preference Assessment Measure, Convenience Subscale (0-4 Points)
Description: as for outcome 39
Time Frame: Baseline
Population: Data available at this time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 74 | 75
units on a scale
  Convenience of Motor Skill Training | 2.65 (0.96) | 2.45 (0.96)
  Convenience of Strength and Flexibility Exercise: number analyzed (Participants) | 73 | 74
  Convenience of Strength and Flexibility Exercise | 3.01 (0.89) | 2.76 (0.93)

43. Other Pre Specified Outcome: Change in Direct and Indirect Health Care Costs (Estimated Costs) From Baseline to Completion of Initial 6 Week Intervention Phase
Description: Background/Purpose: These are measures of costs associated with healthcare over the intervention phase. Procedure: Direct health costs will be estimates of the cost of (1) medication using average wholesale price and wholesale acquisition cost and (2) health services and medical equipment using the Medicare allowable cost. Indirect health costs will be estimated using absenteeism and presenteeism measures.
Time Frame: Baseline, completion of initial 6 week intervention phase
Population: The exploratory economic analyses we proposed to examine direct (medication and health services use and medical equipment) and indirect (absenteeism and presenteeism) health costs are not to be conducted. The decision was based on large budget cuts that limited our ability to financially support the personnel to conduct the analyses
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 0 | 0

44. Other Pre Specified Outcome: Change in Direct and Indirect Healthcare Costs (Estimated Costs) From Completion of Initial 6 Week Intervention Phase to 6 Months After Initial Intervention Phase
Description: Background/Purpose: These are measures of costs associated with healthcare from completion of the initial 6 week intervention phase to 6 months after the initial intervention phase.. Procedure: Direct health costs will be estimates of the cost of (1) medication using average wholesale price and wholesale acquisition cost and (2) health services and medical equipment using the Medicare allowable cost. Indirect health costs will be estimated using absenteeism and presenteeism measures.
Time Frame: Completion of initial 6 week intervention phase, 6 months after initial intervention phase
Population: as for outcome 43
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 0 | 0

45. Other Pre Specified Outcome: Change in Direct and Indirect Healthcare Costs (Estimated Costs) From 6 Months After Initial Intervention Phase to 12 Months After Initial Intervention Phase
Description: Background/Purpose: These are measures of costs associated with healthcare from 6 months after the initial intervention phase to 12 months after the initial intervention phase. Procedure: Direct health costs will be estimates of the cost of (1) medication using average wholesale price and wholesale acquisition cost and (2) health services and medical equipment using the Medicare allowable cost. Indirect health costs will be estimated using absenteeism and presenteeism measures.
Time Frame: 6 months after initial intervention phase, 12 months after initial intervention phase
Population: as for outcome 43
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Study recruitment began in December of 2013 and all study participation ended November of 2017 therefore any adverse event data would be collected between those study time points. Participation for any given individuals was approximately 14 months.
Arm/Group | Motor Skill Training | Strength and Flexibility Exercise
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/75
Serious Adverse Events (participants affected / at risk) | 1/74 | 1/75
Other Adverse Events (participants affected / at risk) | 43/74 | 34/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motor Skill Training (N=74) | Strength and Flexibility Exercise (N=75)
Non-Related to Treatment: Ductal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Specific Adverse Event Terms were not used
Non-Related to Treatment: Disc Herniation Surgery (Surgical and medical procedures) | 0 (0) | 1 (1) — Specific Adverse Event Terms were not used
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Motor Skill Training (N=74) | Strength and Flexibility Exercise (N=75)
Non-Related to Treatment: Worsening of symptoms (Musculoskeletal and connective tissue disorders) | 37 | 25 — An increase in the intensity of low back pain symptoms or peripheralization of symptoms that lasts for greater than 4 hours and has not fully resolved after 24 hours. Not associated with treatment. Systematic assessment during treatment phase.
Related to Treatment: Worsening of symptoms (Musculoskeletal and connective tissue disorders) | 1 | 2 — An increase in the intensity of low back pain symptoms or peripheralization of symptoms that lasts for greater than 4 hours and has not fully resolved after 24 hours. Associated with treatment. Systematic assessment during treatment phase.
Non-Related to Treatment: non-serious (General disorders) | 5 | 7 — Specific Adverse Event Terms were not used

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT02027623/Prot_SAP_000.pdf